CLINICAL TRIAL: NCT06281509
Title: The Potential Relationship Between the Palmaris Longus Muscle Prevalence and Dupuytren Disease: a Comparative Study
Brief Title: Palmaris Longus Muscle and Dupuytren
Acronym: Palmaris
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S68374
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Dupuytren's Disease
MeSH Terms: conditions — Dupuytren Contracture | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Two groups: Patients with Dupuytren Disease and healthy control group. They will be age matched (50 years of age or higher) with the objective to have a proportionate division (50/50) between the genders.
Masking Description: No masking will be done in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with Dupuytren disease (Experimental): 120 individuals diagnosed with Dupuytren disease (primary or recurrent).
  Interventions: Procedure: Non-invasive tests to determine the presence or absence of the palmaris longus tendon in both hands.; Procedure: Ultrasound
- Healthy controls (Experimental): 120 participants with no other medical conditions affecting the function of the hand (musculoskeletal pathology, vascular or neurological conditions such as CRPS, rheumatoid arthritis and paralysis).
  Interventions: Procedure: Non-invasive tests to determine the presence or absence of the palmaris longus tendon in both hands.; Procedure: Ultrasound

INTERVENTIONS:
Procedure: Non-invasive tests to determine the presence or absence of the palmaris longus tendon in both hands. — Schaeffer's test (flexion of the wrist while the pinky and thumb are pressed against each other) Thompson's test (wrist flexion with a clenched fist) Mishra test I (wrist flexion while the examiner pushes the hand back) Mashra test II (thumb opposition while flexing the wrist)
Procedure: Ultrasound — A small mobile ultrasound device will be used to further asses the presence of the tendon.

SUMMARY:
Dupuytren disease is a medical condition characterized by the painless formation of nodules in the palm of the hand. Cords are formed on the palmar fascia, a connective tissue sheet in the palm of the hand. This fascia is seen as the vestigial remnant of the palmaris longus tendon. The PLM attaches to the fascia palmaris. A muscle that not everyone has and can therefore be clearly missed. This raises the question of whether the presence of the musculus palmaris longus has any association with the development, recurrence and/or progression of DD and contractures. To investigate a potential predisposition, this study intend to assess the prevalence of the PLM in a group of individuals affected by DD and compare it with a control group (age matched, no signs of DD) without the condition.

DETAILED DESCRIPTION:
Dupuytren disease is also known as Dupuytren contracture. It is a medical condition characterized by the painless formation of nodules in the palm of the hand. As the disease progresses, approximately 21% - 50% of all patients experience a transformation of these nodules (stage 0/N of Tubiana) into cord-like structures. These cords, in turn, lead to finger contractures (Tubiana stages 1-4) with impairment of hand mobility and stiffening of the palmar skin. The cords are formed on the palmar fascia, a connective tissue sheet in the palm of the hand. This fascia is seen as the vestigial remnant of the palmaris longus tendon. The PLM attaches to the fascia palmaris. A muscle that not everyone has and can therefore be clearly missed. This raises the question of whether the presence of the musculus palmaris longus has any association with the development, recurrence and/or progression of DD and contractures. To investigate a potential predisposition, this study intend to assess the prevalence of the PLM in a group of individuals affected by DD and compare it with a control group (age matched, no signs of DD) without the condition. Interestingly, prior research has already explored this topic. Despite the publication dating back to 1986, it reported a significantly higher occurrence of the palmaris longus tendon in patients affected by DD. Furthermore, a second article from the same year concluded a significant decrease in recurrence when the palmaris longus tendon was resected in combination with regional fasciectomy. Remarkably, no other research on this topic was found despite the promising results of both articles.

ELIGIBILITY:
Inclusion Criteria:

* The participant or his/her legally authorized representative voluntary signed the informed consent prior to the first assessment.
* 50 years of age or higher.
* Has Dupuytren disease (primary or recurrent). (Only applicable for participants of DD group)
* Has no medical conditions affecting the function of the hand (musculoskeletal pathology, vascular or neurological conditions such as CRPS, rheumatoid arthritis and paralysis). (Only applicable for participants of control group)

Exclusion Criteria:

* Patients < 50 years
* Patients with cognitive impairments.
* Patients showing signs of medical conditions affecting the function of the hand (musculoskeletal pathology, vascular or neurological conditions such as CRPS, rheumatoid arthritis and paralysis). (Only applicable for participants of control group)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
PLM in the DD versus control | Baseline
  Percentual prevalence of the Palmaris Longus Muscle in the Dupuytren Disease-group versus the control group.
PML in mild versus severe DD-group | Baseline
  Percentual prevalence of the Palmaris Longus Muscle in the mild (stage 0/N of Tubiana) Dupuytren Disease-group versus the severe (Tubiana stages 1-4) Dupuytren Disease-group.

SECONDARY OUTCOMES:
PLM presence in DD affected group | Baseline
  Percentual prevalence of the Palmaris Longus Muscle in the Dupuytren Disease-group
PLM presence in control group | Baseline
  Percentual prevalence of the Palmaris Longus Muscle in the control group
Dominant versus non-dominant hand | Baseline
  Percentual prevalence of the Palmaris Longus Muscle in the dominant hand versus the non-dominant hand for both Dupuytren Disease-group and control group.
Male versus female population | Baseline
  Percentual prevalence of the Palmaris Longus Muscle in male versus female population.

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Degreef, Prof. Dr., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No